CLINICAL TRIAL: NCT05406401
Title: A Multicenter, Open-label, Phase 2 Dose Escalation and Confirmation, and Efficacy Expansion Study of Zilovertamab Vedotin (MK-2140) in Combination With R-CHP in Participants With DLBCL (waveLINE)
Brief Title: A Study of Zilovertamab Vedotin (MK-2140) in Combination With Cyclophosphamide, Doxorubicin, and Prednisone Plus Rituximab or Rituximab Biosimilar (Truxima) (R-CHP) in Participants With Diffuse Large B-Cell Lymphoma (DLBCL) (MK-2140-007)
Acronym: waveLINE-007
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 2140-007; MK-2140-007 (Other: MSD); 2022-501380-40 (Registry Identifier: EU CT); U1111-1280-2348 (Other: UTN); 2021-005861-41 (EudraCT Number)
Record Dates: First submitted 2022-06-01; First posted 2022-06-06 (Actual); Last update posted 2024-10-15 (Actual); Status verified 2024-10

CONDITIONS: Lymphoma, Large B-Cell, Diffuse (DLBCL)
MeSH Terms: conditions — Lymphoma | interventions — Cyclophosphamide; Doxorubicin; Rituximab; Prednisone; Prednisolone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Zilovertamab Vedotin + R-CHP: Dose Escalation/Confirmation (Experimental): Participants in the dose escalation/confirmation phase receive a dose level of zilovertamab vedotin (from 1.5 mg/Kg up to 2.5 mg/Kg) plus 750 mg/m^2 cyclophosphamide, 50 mg/m^2 doxorubicin, and 375 mg/m^2 rituximab or rituximab biosimilar (truxima) administered by intravenous (IV) infusion on Day 1 of each 21-day cycle (Q3W) for up to 8 cycles (up to approximately 5.5 months). Participants also receive 100 mg prednisone or prednisolone per day during Days 1-5 of each 21-day cycle for up to 8 cycles (up to approximately 5.5 months).
  Interventions: Biological: Zilovertamab Vedotin; Drug: Cyclophosphamide; Drug: Doxorubicin; Biological: Rituximab; Biological: Rituximab Biosimilar; Drug: Prednisone; Drug: Prednisolone
- Zilovertamab Vedotin + R-CHP: Efficacy Expansion (Experimental): Participants in the efficacy expansion phase receive the RP2D of zilovertamab vedotin plus 750 mg/m^2 cyclophosphamide, 50 mg/m^2 doxorubicin, and 375 mg/m^2 rituximab or rituximab biosimilar (truxima) administered by intravenous (IV) infusion on Day 1 of each 21-day cycle (Q3W) for up to 8 cycles (up to approximately 5.5 months). Participants also receive 100 mg prednisone or prednisolone per day during Days 1-5 of each 21-day cycle for up to 8 cycles (up to approximately 5.5 months).
  Interventions: Biological: Zilovertamab Vedotin; Drug: Cyclophosphamide; Drug: Doxorubicin; Biological: Rituximab; Biological: Rituximab Biosimilar; Drug: Prednisone; Drug: Prednisolone

INTERVENTIONS:
Biological: Zilovertamab Vedotin — IV infusion
  Other Names: MK-2140; VLS-101
Drug: Cyclophosphamide — IV infusion
  Other Names: CYTOXAN®; NEOSAR®
Drug: Doxorubicin — IV infusion
  Other Names: ADRIAMYCIN®
Biological: Rituximab — IV infusion
  Other Names: RITUXAN®
Biological: Rituximab Biosimilar — IV infusion
  Other Names: TRUXIMA®
Drug: Prednisone — IV or oral administration (per local guidelines)
Drug: Prednisolone — IV or oral administration (per local guidelines)

SUMMARY:
This study consists of a dose escalation/confirmation phase and an efficacy expansion phase. The dose escalation/confirmation phase is to determine the safety and tolerability and establish a preliminary recommended Phase 2 dose (RP2D) of zilovertamab vedotin when administered in combination with R-CHP in participants with DLBCL who have received no prior treatment for their disease. The efficacy expansion phase is to determine the efficacy of the RP2D of zilovertamab vedotin when administered in combination with R-CHP in participants with DLBCL who have received no prior treatment for their disease.

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion:

* Has histologically confirmed diagnosis of DLBCL by prior biopsy
* Has PET-positive disease verified by blinded independent central review (BICR) at screening, defined as 4-5 on the Lugano response criteria 5-point scale
* Has received no prior treatment for DLBCL
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 assessed within 7 days prior to the start of study intervention

Exclusion:

* Has a history of transformation of indolent disease to DLBCL
* Has received solid organ transplant at any time
* Has received a diagnosis of primary mediastinal B-cell lymphoma (PMBCL)
* Has clinically significant (ie, active) cardiovascular disease: cerebral vascular accident/stroke (<6 months prior to enrollment), myocardial infarction (<6 months prior to enrollment), unstable angina, congestive heart failure (New York Heart Association Classification Class ≥II), or serious cardiac arrhythmia requiring medication
* Has pericardial effusion or clinically significant pleural effusion
* Has ongoing Grade >1 peripheral neuropathy
* Has a demyelinating form of Charcot-Marie-Tooth disease
* History of a second malignancy unless potentially curative treatment has been completed with no evidence of malignancy for 2 years with the exception of participants who underwent successful definitive resection of basal cell carcinoma of the skin, squamous-cell carcinoma of the skin, or carcinoma in situ, excluding carcinoma in situ of the bladder
* Has received prior radiotherapy within 28 days of start of study intervention
* Has ongoing corticosteroid therapy (exceeding 30 mg daily of prednisone equivalent)
* Has received a live or live-attenuated vaccine within 30 days before the first dose of study intervention
* Has received a strong inhibitor or inducer of CYP3A4 (including itraconazole, ketoconazole, posaconazole, or voriconazole) within 7 days prior to the start of study intervention or expected requirement for chronic use of a strong CYP3A4 inhibitor until <30 days after the last dose
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 28 days before the first dose of study intervention
* Has known active central nervous system (CNS) lymphoma
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known active hepatitis C virus infection
* Has a known active hepatitis B virus infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-07-14 (Actual); Primary Completion 2029-04-26 (Estimated); Study Completion 2029-04-26 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Who Experienced Dose-limiting Toxicities (DLTs) in Cycle 1 | Cycle 1 (up to 21 days)
  DLTs will be evaluated using the Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0 and are defined as any drug-related adverse event (AE) observed during the DLT evaluation period (e.g. Cycle 1) that results in a change to a given dose or a delay in initiating the next cycle. The number of participants with DLTs in Cycle 1 will be reported.
Number of Participants Who Experienced At Least One AE | Up to approximately 8 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experience an AE will be reported.
Number of Participants Who Discontinued Study Treatment Due to an AE | Up to approximately 5.5 months
  An AE is any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinue study treatment due to an AE will be reported.
Complete Response Rate (CRR) per Lugano Response Criteria | Up to approximately 60 months
  CRR is defined as the percentage of participants who achieve a Complete Response (CR) per Lugano response criteria [Cheson, B. D., et al 2014] for malignant lymphoma as assessed by the investigator. Assessment includes anatomic imaging with computed tomography (CT) or magnetic resonance imaging (MRI), metabolic imaging with positron emission tomography (PET), and clinical findings including physical examination and bone marrow biopsy results. The percentage of participants with CRR will be reported.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) per Lugano Response Criteria | Up to approximately 60 months
  ORR is defined as the percentage of participants who achieve a CR or PR per Lugano response criteria [Cheson, B. D., et al 2014] for malignant lymphoma as assessed by the investigator. Assessment includes anatomic imaging with CT or MRI, metabolic imaging with PET, and clinical findings including physical examination and bone marrow biopsy results. The percentage of participants with ORR will be reported.
Duration of Response (DOR) per Lugano Response Criteria | Up to approximately 60 months
  For participants who demonstrate a confirmed CR or PR per Lugano response criteria [Cheson, B. D., et al 2014] for malignant lymphoma, DOR is defined as the time from the first documented evidence of CR or PR until disease progression or death due to any cause, whichever occurs first. CR and PR assessment includes anatomic imaging with CT or MRI, metabolic imaging with PET, and clinical findings including physical examination and bone marrow biopsy results. DOR as assessed by the investigator will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (22):
- Canada (3):
  - BC Cancer Victoria-Clinical Trials Unit ( Site 0105), Victoria, British Columbia
  - William Osler Health System ( Site 0106), Toronto, Ontario
  - Hopital du Sacre-Coeur de Montreal ( Site 0108), Montreal, Quebec
- Israel (2):
  - Hadassah Medical Center ( Site 0401), Jerusalem
  - Sheba Medical Center-Hemato Oncology ( Site 0400), Ramat Gan
- Italy (5):
  - Fondazione Policlinico Universitario Agostino Gemelli-ISTITUTO DI EMATOLOGIA ( Site 0306), Rome, Lazio
  - Ospedale San Raffaele-Unità Linfomi ( Site 0305), Milan, Lombardy
  - Az. Osp. Ospedali Riuniti VILLA SOFIA-CERVELLO-EMATOLOGIA I ( Site 0307), Palermo, Sicily
  - Azienda Ospedaliera Universitaria Careggi-SOD Ematologia ( Site 0308), Florence, Tuscany
  - Azienda Ospedaliera Nazionale SS. Antonio e Biagio e Cesare -Azienda Ospedaliera Nazionale SS. Ant, Alessandria
- Poland (4):
  - Narodowy Instytut Onkologii im. Marii Sklodowskiej-Curie - P-Kilinka Onkologii I Hematologii ( Site, Warsaw, Masovian Voivodeship
  - Uniwersyteckie Centrum Kliniczne-Klinika Hematologii i Transplantologii ( Site 0504), Gdansk, Pomeranian Voivodeship
  - Narodowy Instytut Onkologii - Oddzial w Gliwicach ( Site 0505), Gliwice, Silesian Voivodeship
  - Wojewodzkie Wielospecjalistyczne Centrum Onkologii i Traumat-Oddiał Hematologii Ogólnej ( Site 0503), Lodz, Łódź Voivodeship
- South Korea (2):
  - Seoul National University Hospital ( Site 0201), Seoul
  - Samsung Medical Center ( Site 0200), Seoul
- Spain (3):
  - HOSPITAL UNIVERSITARIO VIRGEN DEL ROCIO-Hematology ( Site 0704), Seville, Andalusia
  - Instituto Catalan de Oncologia - Hospital Duran i Reynals-Haematology Department ( Site 0703), L'Hospitalet Del Llobregat, Barcelona
  - Hospital Universitario Fundación Jiménez Díaz-Oncology & Hematology ( Site 0700), Madrid
- Turkey (Türkiye) (3):
  - Mega Medipol-Hematology ( Site 0808), Stanbul, Istanbul
  - Ankara Universitesi Tip Fakultesi Hastanesi-hematology ( Site 0801), Ankara
  - Trakya University ( Site 0805), Edirne

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26131&tenant=MT_MSD_9011